CLINICAL TRIAL: NCT04915248
Title: An Open Label, Phase 2 Study to Evaluate Activity and Safety of Daratumumab in Combination With Bortezomib and Dexamethasone in Patients With Relapsed or Refractory Plasmablastic Lymphoma (DALYA Trial)
Brief Title: Study to Evaluate Combined Treatment of Daratumumab, Bortezomib and Dexamethasone in PBL Patients.
Acronym: FIL_DALYA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_DALYA
Record Dates: First submitted 2021-05-14; First posted 2021-06-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Plasmablastic Lymphoma
Keywords: Relapsed; Refractory; Plasmablastic; lymphoma; PBL; Daratumumab; Bortezomib; Dexamethasone
MeSH Terms: conditions — Plasmablastic Lymphoma; Recurrence; Lymphoma | interventions — daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients registered in the DALYA trial (Experimental): Treatment consists of an induction phase (every 21 days) planning one course (cycle 1) of daratumumab as single agent followed by 8 courses (cycles 2-9) of daratumumab in combination with bortezomib and dexamethasone (DVd regimen).
  Patients achieving at least a SD after induction will be addressed to the maintenance phase (every 28 days), planning a maximum of 6 cycles (cycles 10-15) of daratumumab as single agent until disease progression, unacceptable toxicity, withdrawal of consent and/or the investigator decision.
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Induction phase planning one course (cycle 1) of daratumumab as single agent followed by 8 courses (cycles 2-9) of daratumumab in combination with bortezomib and dexamethasone (DVd regimen).
  Patients achieving at least a SD after induction will be addressed to the maintenance phase, planning a maximum of 6 cycles (cycles 10-15) of daratumumab as single agent.
  Other Names: Daratumumab sc
Drug: Bortezomib — Induction phase planning one course (cycle 1) of daratumumab as single agent followed by 8 courses (cycles 2-9) of daratumumab in combination with bortezomib and dexamethasone (DVd regimen).
  Patients achieving at least a SD after induction will be addressed to the maintenance phase, planning a maximum of 6 cycles (cycles 10-15) of daratumumab as single agent.
  Other Names: Bortezomib sc
Drug: Dexamethasone — Induction phase planning one course (cycle 1) of daratumumab as single agent followed by 8 courses (cycles 2-9) of daratumumab in combination with bortezomib and dexamethasone (DVd regimen).
  Patients achieving at least a SD after induction will be addressed to the maintenance phase, planning a maximum of 6 cycles (cycles 10-15) of daratumumab as single agent.
  Other Names: Dexamethasone os

SUMMARY:
It is an open-label, multicenter, phase II, single arm trial to Evaluate Activity and Safety of Daratumumab in combination with Bortezomib and Dexamethasone in patients about 28 patients with Relapsed or Refractory Plasmablastic lymphoma.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase II, single arm trial. Patients will be recruited over 18 months in 19 FIL centers and it is expected that a total of 28 patients will start treatment. Analysis of the primary endpoint of the study is planned approximately after 12 months from the enrollment of the last patient, regardless of the response to protocol treatment of this patient. The total duration of the study is 30 months (~2.5 years).

Patients will be enrolled based on the local diagnosis and the local assessment of CD38 expression ≥ 5%. The screening phase of the study includes baseline assessments according to local practice and those required by the study.

Samples coming from the most recent biopsy, and if available also those used for the first diagnosis, are to be collected and sent afterwards, upon request of the FIL Offices, to one of the three FIL designed central laboratories. Central diagnosis review and CD38 assessment will be performed during or at the end of the study conductance; there's no need to wait for central results to start protocol treatment.

Protocol treatment consists of an induction phase planning one course (cycle 1) of daratumumab sc as single agent followed by 8 courses (cycles 2-9) of daratumumab sc in combination with bortezomib sc and dexamethasone (DVd regimen).

Patients achieving at least a SD after induction will be addressed to the maintenance phase, planning a maximum of 6 cycles (cycles 10-15) of daratumumab sc as single agent.

Induction cycles will be administered every 21 days, while maintenance cycles will be administered every 28 days.

Treatment with DVd or daratumumab single agent will be discontinued before completion of planned cycles in case of disease progression, unacceptable toxicity, withdrawal of consent and/or the investigator determines that further therapy is not in the patient best interest (e.g., due to non-compliance, toxicity, etc.). Adverse events according to CTCAE will be monitored from the first dose of induction treatment, throughout maintenance phase and for 30 days after the last dose of protocol treatment with the study drug or 30 days after the last dose of drug in case of early discontinuation from any cause.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed plasmablastic lymphoma according to WHO 2017, CD38-positive by immunohistochemistry (≥5% of positive cells) Local diagnosis of PBL and local CD38 assessment ≥5% will suffice for enrollment and start of treatment.
2. Patients with plasmablastic lymphoma relapsed or refractory:

   * after at least one line of conventional-dose chemotherapy followed or not by autologous stem cell transplantation;
   * after at least one line of conventional-dose chemotherapy and not eligible for salvage autologous or allogeneic transplantation;
3. ECOG Performance Status ≤ 3;
4. Age ≥ 18 years;
5. Both HIV-negative and HIV-positive patients are eligible;
6. HIV infection responsive to ongoing cART (combination antiretroviral therapy);
7. At least one measurable disease lesion identifiable by imaging:

   * A nodal lesion must be at least 11 mm x 11 mm OR ≥ 16 mm in the greatest transverse diameter (regardless of short axis measurement).
   * An extranodal lesion must be at least 10 mm x 10 mm.
8. Women of childbearing potential (WOCBP) and men must agree to use effective contraception if sexually active. This applies for the time period between signing of the informed consent form and 7 months (for women) o 4 months (for men) after last administration of bortezomib or 6 months after last daratumumab dose, regardless of sex. A woman is considered of childbearing potential, i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control method (failure rate of less than 1%) e.g., intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, and sexual abstinence. The use of condoms by male patients is required unless the female partner is permanently sterile.

   WOCBP must have two negative pregnancy tests as verified by the study doctor prior to starting study therapy and must agree to undergo monthly pregnancy testing during the course of the study and after end of study therapy if clinically indicated. This applies even if the subject practices complete abstinence from heterosexual contact.
9. Subject understands and voluntarily signs and dates an informed consent form approved by an Independent Ethics Committee (IEC), prior to the initiation of any screening or study-specific procedures
10. Subject must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Histologic diagnosis different from confirmed plasmablastic lymphoma according to WHO 2017 and/or CD38 expression < 5% of positive cells
2. CNS involvement
3. Patients with known hypersensitivity to the investigational drug or to product components or severe allergic or anaphylactic reactions to humanized products
4. Subject has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, investigational therapy including targeted small molecule agents within 14 days prior to the first dose of study drug
5. Concomitant Kaposi sarcoma; however, patients with only skin involvement of KS can be included.
6. Subject is:

   * Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]. Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [HBcAb] ± antibodies to hepatitis B surface antigen [HBsAb]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (HBsAb positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
   * Known to be seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)
7. Any history of another cancer during the last 5 years with the exception of non-melanoma skin tumors, in situ cervical carcinoma, or in situ breast cancer treated with curative intent with no history of metastatic disease.
8. Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis or tuberculosis. Drugs for HIV treatment are allowed, as per local investigator prescription.
9. Active ongoing infection from SARS-CoV-2.
10. Screening laboratory values (due to causes different than lymphoma):

    * Absolute neutrophil count (ANC) <1.0 x 109/L (unless secondary to documented marrow involvement by lymphoma)
    * Platelet count <75 x 109/L
    * Hemoglobin < 7.5 g/dL
    * Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) > 3.5 times the upper limit of normal (ULN)
    * Alkaline phosphatase > 3.5 times ULN
    * Bilirubin > 2 times x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
    * Serum Creatinine Clearance < 20 ml/h
11. Subject has clinically significant cardiac disease, including:

    * Myocardial infarction within 6 months before date of registration, or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
    * Cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] current version Grade 2 or higher) or clinically significant ECG abnormalities. Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) > 470 msec
12. Evidence of any other clinically significant uncontrolled condition(s)
13. Significant history of neurologic, psychiatric, endocrinological, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent
14. Breastfeeding women or women with a positive pregnancy test at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 30 months
  Response assessment will be done at each restaging. The best overall response will be defined as the best response between the date of beginning of therapy and the last response evaluation. Patients without response assessment (due to whatever reason) will be considered as non-responders.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 30 months
  From the date of starting therapy and the date of disease progression, relapse or death from any cause. Responding patients according to the Lugano classification response Criteria and patients who are lost to follow-up will be censored at their last assessment date.
Overall survival (OS) | 30 months
  From the date of starting therapy and the date of death from any cause. Patients alive and those who are lost to follow-up at the time of the final analysis will be censored at the date of the last contact.
Duration of response (DOR) | 30 months
  For all patients who achieved a response (CR or PR) according to Response Criteria for NHL with PET (Lugano 2014) and it is measured from the date when criteria for response are met (CR or PR) until the date of progression (including death due to progression) or relapse. Patients without relapse or progression or with death from other cause than progression will be censored at their last assessment date.
Number of participants with treatment-related adverse events as assessed by current version of CTCAE. | 30 months
  The safety of daratumumab as single agent and in combination with bortezomib/dexamethasone will be assessed in all patients who have received at least one dose of study medication. Rates of adverse events and of serious adverse events will be will be presented with two sided 95% confidence intervals.
Rate of Complete Remission (CRR) | 30 months
  Comparison of ORR and CRR before and after maintenance, and by evaluation of rate of conversion of SD to PR and of SD/PR to CR with daratumumab maintenance.
Relationship between CD38 expression on lymphoma cells, assessed by immunohistochemistry, and the response rate. | 30 months
  The extent of CD38 expression evaluated by immunochemistry on the diagnostic biopsy-tissue will be correlated with response measured according to the Lugano 2014 criteria at various timepoints: after induction cycle 1, after induction cycles 3, 6 and 9 (end of induction, EOI); after maintenance cycles 12 and 15 (end of treatment, EOT). correlated with response measured according to the Lugano 2014 criteria at various endpoints.
Impact of daratumumab and bortezomib treatment on biological cell profiles. | 30 months
  The impact of daratumumab and bortezomib treatment in immune activation (CD38, CD25, HLA-DR), T cell differentiation (naïve, central memory, effector memory and terminal effector memory T cell subset) and on circulating myeloid-derived suppressor cells (MDSC) as well as Treg will be evaluated by multiparametric flow cytometry (84 multiple staining). Peripheral blood samples will be collected in different timepoints: before treatment start; after cycle 1; after cycle 3 and at EOT.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Ferreri, Dr., Principal Investigator — Unità Linfomi - Dipartimento Oncoematologia -Istituto Scientifico San Raffaele - Milano
Locations (18):
- Italy (18):
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona, Ancona
  - Aviano - IRCCS Centro di Riferimento Oncologico di Aviano - Divisione di Oncologia e dei Tumori immuto-correlati, Aviano
  - A.O. Spedali Civili di Brescia - Ematologia, Brescia
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - Milano - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Miano
  - Istituto Scientifico San Raffaele, Unità Linfomi - Dipartimento Oncoematologia, Milan
  - Monza - ASST MONZA Ospedale S. Gerardo - Ematologia, Monza
  - Napoli - AORN - Azienda Ospedaliera dei Colli Monald - U.O.C. Oncologia, Napoli
  - U.O. Ematologia AO di Padova, Padua
  - A.O. Universitaria Policlinico Giaccone Di Palermo, Palermo
  - Ematologia IRCCS Policlinico S. Matteo di Pavia, Pavia
  - AO Arcispedale S.Maria Nuova Ematologia, Reggio Emilia
  - Roma - IRCCS Spallanzani - Servizio di Ematologia in malattie infettive, Roma
  - Roma - Ospedale S. Camillo - Ematologia, Roma
  - A.O. S. Maria di Terni - S.C. Oncoematologia, Terni
  - A.O. Universitaria Citta' Della Salute E Della Scienza Di Torino, Torino
  - Struttura Complessa di Ematologia PO TREVISO, Treviso
  - AOU Integrata di Verona - U.O. Ematologia, Verona

IPD SHARING:
Plan to Share IPD: No